CLINICAL TRIAL: NCT06580808
Title: Effects of Inspiratory Muscle Training in Children After Fontan Surgery.
Brief Title: Inspiratory Training in Children After Fontan
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Sao Paulo General Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 38501214.8.0000.0068
Record Dates: First submitted 2024-08-16; First posted 2024-08-30 (Actual); Last update posted 2024-08-30 (Actual); Status verified 2017-09

CONDITIONS: Respiratory Muscle Weakness
Keywords: congenital heart disease; Fontan procedure; rehabilitation; physiotherapy; inspiratory muscle training
MeSH Terms: conditions — Heart Defects, Congenital

STUDY DESIGN:
Intervention Model Description: Patients in the Fontan group were randomized into the Fontan Training Group (FTG) and Fontan Control Group. The FTG performed inspiratory muscle training with the Power Breth device with an initial load of 40% of the maximum inspiratory pressure obtained by measuring the maximum inspiratory pressure by manovacuometry. The training lasted 2 months. The patient was asked to perform the training every day with 3 series of 20 breaths. The training was monitored in person and remotely by videoconference; the load was increased gradually when it was perceived that it was already easy or reported by the child.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Control Group (No Intervention): The control group consisted of 18 healthy children. These children underwent cardiopulmonary testing, spirometry, chest ultrasound to assess the diaphragm, 6-minute walk test, respiratory muscle strength and quality of life. These tests were performed to assess the results of these tests in patients without previous illnesses.
- Fontan Training Group (Active Comparator): The Fonta training group consisted of 14 children in the late postoperative period of Fontan surgery. These children underwent cardiopulmonary testing, spirometry, chest ultrasound to assess the diaphragm, 6-minute walk test, respiratory muscle strength and quality of life. These tests were performed at the initial stage and after two months of inspiratory muscle training to assess the results of these in postoperative patients and what changes the training could bring. The training was performed with the Power Breath device, the carda was quantified at 40% of the force exerted at maximum inspiratory pressure by manovacuometry. The patient was asked to perform 3 sets of 20 repetitions twice over the course of 7 days of the week. Monitoring was done in person and virtually, and the carda was increased according to the evaluator's perception of the ease of the exercise or if the patient reported it to be easy. The training lasted 2 months.
  Interventions: Other: Fontan Training Group
- Fonta Control Group (No Intervention): The Fonta Control Group consisted of 13 children in the late postoperative period of Fontan surgery. These children underwent cardiopulmonary testing, spirometry, chest ultrasound to assess the diaphragm, 6-minute walk test, respiratory muscle strength and quality of life. These tests were performed at the initial stage and after two months to assess the results of these tests in postoperative patients and whether there was any normal behavior.

INTERVENTIONS:
Other: Fontan Training Group — The Fonta training group consisted of 14 children in the late postoperative period of Fontan surgery. These children underwent cardiopulmonary testing, spirometry, chest ultrasound to assess the diaphragm, 6-minute walk test, respiratory muscle strength and quality of life. These tests were performed at the initial stage and after two months of inspiratory muscle training to assess the results of these in postoperative patients and what changes the training could bring. The training was performed with the Power Breath device, the carda was quantified at 40% of the force exerted at maximum inspiratory pressure by manovacuometry. The patient was asked to perform 3 sets of 20 repetitions twice over the course of 7 days of the week. Monitoring was done in person and virtually, and the carda was increased according to the evaluator's perception of the ease of the exercise or if the patient reported it to be easy. The training lasted 2 months.
  Arms: Fontan Training Group

SUMMARY:
This study will assess physical and respiratory capacity, diaphragmatic mobility and quality of life. Healthy children and children who have undergone Fontan surgery will participate. Some children in the late postoperative period of Fontan surgery will be randomized to a group of inspiratory muscle training that will last for 2 months. Children after Fontan surgery will be evaluated twice, once at the beginning and again after two months of follow-up.

DETAILED DESCRIPTION:
This study aims to evaluate physical capacity through cardiopulmonary testing, submaximal physical capacity testing by the 6-minute walk test, respiratory capacity by spirometry, respiratory muscle strength by manovacuometry, diaphragmatic mobility by ultrasound, quality of life by the AUQEI questionnaire. There are three groups, a healthy control group, a Fontan control group and a Fontan intervention group. The intervention will be done by respiratory muscle training using the Power Breath device.

ELIGIBILITY:
Inclusion Criteria:

* Age 8 to 12 years;
* Both sexes;
* No history of other heart disease;
* No history of lung and musculoskeletal diseases;
* >1 year post-operative Fontan Surgery;
* Clinically stable;
* Absence of serious arrhythmias;
* Medical clearance to participate in the study; The legal guardian has agreed to participate in the research and the child has consented

Exclusion Criteria:

* Musculoskeletal alterations;
* Patients with neurological sequelae;
* Patients with genetic syndromes associated with cognitive or psychiatric disorders;
* History of perioperative arrhythmias;
* Patients with uncontrolled heart failure;
* Recent angina;
* Severe arrhythmia;
* Hemoptysis;
* Pulmonary hypertension;
* Diaphragmatic plication;
* Moderate to severe asthma.

Ages: 8 Years to 12 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 45 (Actual)
Dates: Start 2017-09-27 (Actual); Primary Completion 2024-01-13 (Actual); Study Completion 2024-06-10 (Actual)

PRIMARY OUTCOMES:
Assessment of the diaphragm muscle | Baseline to 2 months
  The mobility and thickness of the diaphragm muscle were assessed using ultrasound in M mode. Both variables were analyzed during spontaneous, relaxed breathing in terms of both tidal volume and deep breathing at vital capacity. Muscle mobility was examined along the right and left mid-axillary and parasternal lines with volunteers in both the supine and sitting positions. Muscle thickness was measured while the patients were in the supine position along the mid-axillary lines during both natural, relaxed and deep breathing. Measurements were taken in centimeters, with the largest value selected from at least three reproducible measurements.

SECONDARY OUTCOMES:
Respiratory muscle strength | Baseline to 2 months
  Respiratory muscle strength was measured using maximum inspiratory pressure (MIP) and maximum expiratory pressure (MEP) with a digital manometer calibrated beforehand. The MIP was determined by the maximal inspiratory effort from the residual volume (RV), and the MEP was determined by the maximal expiratory effort from the total lung capacity (TLC). At least three reproducible maneuvers were performed, with the largest value used unless it did not exceed the previous value by more than 20%.
Lung function test | Baseline to 2 months
  Pulmonary volume and capacity were evaluated using the spirometer protocol as recommended by the American Thoracic Society guidelines. For spirometry, at least three acceptable and reproducible maneuvers at each stage were performed using encouragement and positive reinforcement to obtain maximum values. Forced vital capacity (FVC), forced expiratory volume in one second (FEV1), and the FEV1/FVC ratio were studied, and the predicted values were calculated from previously reported equations
Six-minute walk test | Baseline to 2 months
  A submaximal analysis of physical capacity was conducted using the six-minute walk test (6MWT), following the protocol of the American Thoracic Society[16]. The patients were instructed to walk as quickly as possible without running for six minutes, while the distance covered was recorded. Breaks during the walk were allowed if needed. The data analyzed included the distance covered in meters, heart rate, respiratory rate, peripheral oxygen saturation, blood pressure, and the Modified Borg Scale for Fatigue. These measurements were taken at rest one minute before the test, immediately after the test, two minutes after the test if there was an interruption, and five minutes after the test.
Change in quality of life measurement | Baseline to 2 months
  The evaluation of quality of life was conducted using the Self-imaginary Questionnaire on Children's Quality of Life (Autoquestionnaire Qualité de Vie Enfant Imagé). This scale consists of closed questions about the point of view for children aged 4 to 12 years, and their answers are directed toward 'very happy', 'happy', 'unhappy', or 'very unhappy', supported by an image of a child in these emotional states. The survey included 26 analysis items related to socialization, family relationships, activities, health, isolation, and other functions. The items were divided into factors such as autonomy, leisure, functions, family, and the legal value of the answers. The sum of all the questions generates a score with a maximum of 78. Scores less than 48 are considered to indicate a loss in quality of life. The questionnaire was validated and translated by Assumpçao et al.
Improvement exercise tolerance and functional capacity (peak VO2) | Baseline to 2 months
  Change in functional capacity will be performed by cardiopulmonary exercise test and will be expressed by Peak VO2 and Predicted Peak VO2 (%). After the training program, an increase in the peak VO2(mL/kg/min) value between 10 to 15% is expected in relation to the baseline value.

CONTACTS AND LOCATIONS:
Overall Officials: Marcelo B Jatene, Manager, Study Director — Heart Institute, University of São Paulo; Joao Bruno PD Silveira, Execution, Principal Investigator — Heart Institute, University of São Paulo
Locations (1):
- Heart Intitute, São Paulo, Brazil

IPD SHARING:
Plan to Share IPD: Yes
If any researcher has any questions about the research or wants to replicate it, I am available to clarify them. If any agency or entity has any questions about the results, they can be made available based on their confidentiality and ethical responsibility to be reanalyzed and reproduced.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: The data will be available for possible checks at any time from now on.
Access Criteria: To access the data, if necessary, simply make a formal request and describe the reason for doing so.